CLINICAL TRIAL: NCT02654457
Title: Identification and Semi-Quantification of Ki-67 Protein Expression Status in Formalin Fixed, Paraffin-embedded Normal and Neoplastic Breast Tissue
Brief Title: Identification and Semi-Quantification of Ki-67 Protein Expression Status
Status: Completed | Type: Observational
Sponsor: Applied Spectral Imaging Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: ASI-Ki-67-IHC
Record Dates: First submitted 2015-02-05; First posted 2016-01-13 (Estimated); Last update posted 2016-01-13 (Estimated); Status verified 2016-01

CONDITIONS: Breast Cancer
Keywords: Immunohistochemical; Ki-67; Breast cancer; IHC
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Women with Breast Cancer #1: IVD Study
  Interventions: Procedure: Women with Breast Cancer
- Women with Breast Cancer #2: IVD Study
  Interventions: Procedure: Women with Breast Cancer
- Women with Breast Cancer #3: IVD Study
  Interventions: Procedure: Women with Breast Cancer

INTERVENTIONS:
Procedure: Women with Breast Cancer — IVD Study

SUMMARY:
The purpose of the study is the identification and semi-quantification of Ki-67 protein expression level in breast cancer tissues by the GenASIs GoPth system as compared to manual reading of the same slides.

The imaging system is intended for diagnostic use as an aid to the pathologist in the detection, counting and classifying ER/PR IHC stained samples

DETAILED DESCRIPTION:
The anti Ki-67 is a semi-quantitative immunohistochemical (IHC) assay to identify the Ki-67 protein expressions in formalin-fixed, paraffin-embedded human breast cancer tissue specimens. Results from the Ki-67 test is indicated as an aid in the assessment of the protein status of breast cancer patients. While the p53 kit provides the antibody that offer direct visualization and semi-quantification of the protein expression through a brightfield microscope, the GenASIs GoPath system is designed to complement the routine workflow of the pathologist in the analysis and review of immunohistochemically stained histologic slides.

ELIGIBILITY:
Inclusion Criteria:

* Slides with nuclear borders of tumor nuclei that is distinguishable, and having good integrity.

Exclusion Criteria:

* Slides that have lots of background that interfere with the analysis

Ages: 21 Years to 89 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women having breast cancer aged 21 and up
Sampling Method: Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2013-12; Primary Completion 2014-05 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
IVD study of Ki67 IHC samples: Accuracy of analysis | 1 Day
  Comparison tests (accuracy) between manual and automatic analysis of antibody expressions. The results from the automatic counting from the clinical studies will be compared to the manual counting analysis.
  Accuracy of the study will be declared "Success" if Positive, Negative and Overall agreement with manual count of the Ki67 antibody at least 85%.
IVD study of Ki67 IHC samples: Repeatability & Reproducibility of analysis | 1 Day
  Repeatability & Reproducibility tests of system analysis of antibody expressions. R&R acceptance criteria of Ki67 are related to the average agreement for between runs, between days and between systems R&R part of the study will be declared "Success" if Positive and Negative average agreement will be at least 80%.